CLINICAL TRIAL: NCT03487003
Title: Comparison of the Clinical Performances of Flexible Laryngeal Mask Airway in Pediatric Patients Under General Anesthesia With or Without Muscle Relaxant: a Randomized Controlled Non-inferiority Trial
Brief Title: Muscle Relaxants on Efficacy of LMA Insertion
Acronym: LMA_MR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Kim, Assistant professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DCMC#3
Record Dates: First submitted 2018-03-15; First posted 2018-04-03 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia Intubation Complication
Keywords: laryngeal mask airway; children, preschool; muscle relaxant
MeSH Terms: conditions — Muscle Hypotonia | interventions — Rocuronium; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized parallel prospective non-inferiority study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MR group (Active Comparator): When the patients asleep, 0.3 mg/kg rocuronium is administered.
  Interventions: Drug: rocuronium
- NMR group (Experimental): When the patients asleep, 0.3 mg/kg saline is administered.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: rocuronium — After standard anesthetic monitoring (non-invasive blood pressure monitor, pulse oximetry, 3-lead echocardiography), patients are inhaled with sevoflurane. When the patients asleep, 0.3 mg/kg rocuronium is administered. After 2 min, flexible laryngeal mask airway (fLMA) is inserted using standard method. The fLMA is inflated with air to 40 cmH2O using manometry. The oropharyngeal leak pressure (OLP) was determined by the method described by Lopez-Gil and colleagues.
  Other Names: Rocuronium bromide
  Arms: MR group
Drug: saline — After standard anesthetic monitoring (non-invasive blood pressure monitor, pulse oximetry, 3-lead echocardiography), patients are inhaled with sevoflurane. When the patients asleep, 0.3 mg/kg saline is administered. After 2 min, flexible laryngeal mask airway (fLMA) is inserted using standard method. The fLMA is inflated with air to 40 cmH2O using manometry. The oropharyngeal leak pressure (OLP) was determined by the method described by Lopez-Gil and colleagues
  Other Names: 0.9% normal saline
  Arms: NMR group

SUMMARY:
The use of laryngeal mask airway (LMA) is increasing in pediatric anesthesia because it provides lesser direct mechanical stimulation of the airway due to being placed above the larynx. However, LMA insertion can be more difficult in children than in adults due to their unique characteristics of pediatric airway. Neuromuscular blocking agents, so-called, muscle relaxants have long been used to facilitate insertion of airway devices. But there are pros and cons for the efficacy of muscle relaxants in LMA insertion, and most studies were investigated in adults.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 7 years of American Society of Anesthesiologists physical status (ASA PS) I or II who are planned to receive ophthalmic surgery under general anesthesia

Exclusion Criteria:

* Refusal of consent
* Present URI or other respiratory symptoms
* Oro or facial anomaly
* Poor dental condition
* who cannot open their mouth or limited mouth opening
* when the tracheal intubation is definitely needed

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure (OLP) | During 1 min after successful LMA intubation
  It was determined by the method describe by Lopez-Gil and colleagues. Briefly, it was measured by closing the expiratory valve of the circle system at a fixed gas flow of 3l/min, recording the airway pressure at which audible leak sound was heard.

SECONDARY OUTCOMES:
Intubation time | During 5-10 min after inhalation of sevoflurane
  from the time of mouth opening until the time at square-wave capnography was detected
Ease of intubation/mask bagging | During 5-10 min after inhalation of sevoflurane
  After successful LMA insertion, investigator recorded subjective difficulty during whole period of LMA manipulation by Likert scale: 1, easy 2, moderate, and 3: difficult.
Fiberoptic view of LMA | During 5min after successful LMA insertion
  The fibreoptic view was assessed by fibreoptic bronchoscopy through the LMA and graded.
Mean blood pressure | During 5-10 min after inhalation of sevoflurane
  mean blood pressure (mmHg) is recorded before and after the insertion of LMA.
Heart rate | During 5-10 min after inhalation of sevoflurane
  Heart rate is (beat per minutes) recorded before and after the insertion of LMA.
Watcha scale every 10 min from time to PACU admission to discharge | During 60 minutes after PACU admission
  On arrival and every 10 min after PACU admission, patients were checked Watcha scale as following 4-point scale
  1. calm
  2. crying, but can be consoled
  3. Crying, cannot be consoled
  4. Agitated and thrashing around
FLACC score on initial, 10, 20, and 30 min | During 60 minutes after PACU admission
  Face, legs, activity, cry, and consolability (FLACC) score is checked every 10min after PACU admission
Eye opening time | During 1 hour after operation
  defined as the interval from the cessation of anesthetics to eye opening
Extubation time | During 1 hour after operation
  time from discontinuation of anesthetics to extubation
Peak inspiratory pressure before and after the surgery | During 4 hour after anesthetic inhalation
  check the peak inspiratory pressure (cmH2O) before and at the end of surgery
Tidal volume ratio before and after the surgery | During 4 hour after anesthetic inhalation
  check the expiratory tidal volume/setting tidal volume ratio before and at the end of surgery
Respiratory adverse events | During 1 hour after operation
  check the adverse events during emergence and PACU stay such as coughing, laryngospasm, bronchospasm, postoperative stridor and mild desaturation; SpO2 <95%.
Postoperative complications | During 1 hour after operation
  check the adverse events including respiratory adverse events, gastric insufflation, excessive secretion, postoperative nausea and vomiting, sore throat, and tinged blood on LMA surface.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kim, MD, PhD, Study Chair — Assistant professor
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gong YH, Yi J, Zhang Q, Xu L. Effect of low dose rocuronium in preventing ventilation leak for flexible laryngeal mask airway during radical mastectomy. Int J Clin Exp Med. 2015 Aug 15;8(8):13616-21. eCollection 2015. PMID 26550303
- [Background] von Ungern-Sternberg BS, Boda K, Chambers NA, Rebmann C, Johnson C, Sly PD, Habre W. Risk assessment for respiratory complications in paediatric anaesthesia: a prospective cohort study. Lancet. 2010 Sep 4;376(9743):773-83. doi: 10.1016/S0140-6736(10)61193-2. PMID 20816545
- [Background] Ghai B, Wig J. Comparison of different techniques of laryngeal mask placement in children. Curr Opin Anaesthesiol. 2009 Jun;22(3):400-4. doi: 10.1097/aco.0b013e3283294d06. PMID 19434792
- [Background] Hattori K, Komasawa N, Miyazaki Y, Kido H, Deguchi S, Minami T. Muscle relaxant facilitates i-gel insertion by novice doctors: A prospective randomized controlled trial. J Clin Anesth. 2016 Sep;33:218-22. doi: 10.1016/j.jclinane.2016.03.058. Epub 2016 May 4. PMID 27555168
- [Background] Chen BZ, Tan L, Zhang L, Shang YC. Is muscle relaxant necessary in patients undergoing laparoscopic gynecological surgery with a ProSeal LMA? J Clin Anesth. 2013 Feb;25(1):32-5. doi: 10.1016/j.jclinane.2012.06.004. Epub 2012 Nov 2. PMID 23122973
- [Derived] Byun SH, Kim SJ, Kim E. Comparison of the clinical performance of the flexible laryngeal mask airway in pediatric patients under general anesthesia with or without a muscle relaxant: study protocol for a randomized controlled trial. Trials. 2019 Jan 9;20(1):31. doi: 10.1186/s13063-018-3141-2. PMID 30626406